CLINICAL TRIAL: NCT00324792
Title: Effect of an Intensive Insulin Therapy on the Production of LTE4 in Patients With Diabetes
Brief Title: I3LTE4: Intensive Insulin Therapy and Production of LTE4 in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DCIC 05 54
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Diabetes Mellitus; Leucotrienes
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Drug: intensive insulin therapy

SUMMARY:
The primary objective of the study is to assess the effect of a 3-month intensive insulin therapy on urinary leukotriene E4 (LTE4) excretion in patients with diabetes.

DETAILED DESCRIPTION:
Our group has recently reported the results of a preliminary cross-sectional study, which demonstrated that the urinary LTE4 excretion is increased in patients with type 1 diabetes. With regard to recent human genetic studies showing that polymorphisms in the 5-lipoxygenase (5-LO) promoter and FLAP haplotypes is linked to cardiovascular disease susceptibility our data suggested the potential interest of LTE4 as a non-invasive biomarker of cardiovascular risk. In diabetes mellitus, further studies are required to evaluate the 5-LO pathway after improvement of glucose control and concomitantly with established inflammatory cardiovascular biomarkers.

The secondary objectives are:

Before and after 3-month intensive insulin therapy- Relationship between a marker of platelet activation (urinary 11-dehydro-thromboxan B2 :11-dehydroTXB2) and urinary LTE4- Relationship between inflammatory plasma markers of cardiovascular risk (hs-CRP and fibrinogen) and urinary LTE4- Relationship between a plasma marker of endothelial dysfunction (sICAM-1) and urinary LTE4- Changes in LTE4 according to patient subgroups (patients with type 1 and type 2 diabetes mellitus)

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus (type 1 or type 2)
* > 18 year-old
* subject has given free, informed written consent
* subject entitled to health insurance cover
* medical follow-up at the department of Diabetology, Grenoble University Hospital
* inappropriate glucose control (HbA1c > 8.5%) requiring an initiation, or revision, of insulin therapy

Exclusion Criteria:

* legal incapacity or limited legal competence
* pregnant women
* heart failure
* impaired renal function,defined by a creatinin clearance < 60 ml/mn according to Cockroft formula
* asthma
* respiratory failure
* IV, IM, SC or oral treatment with cortico-steroids for the last 2 months prior to baseline
* current smoking > cigarettes / day
* any infectious disease for the last 2 months prior to baseline
* baseline CRP > 20 mg/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-05; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
changes in urinary LTE4 excretion and HbA1c after 3-month intensive insulin therapy versus baseline

SECONDARY OUTCOMES:
urinary 11-dehydroTXB2
hs-CRP
fibrinogen
sICAM-1 plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Robert Boizel, Dr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Département d'urologie, néphrologie et endocrinologie-University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Hardy G, Boizel R, Bessard J, Cracowski JL, Bessard G, Halimi S, Stanke-Labesque F. Urinary leukotriene E4 excretion is increased in type 1 diabetic patients: a quantification by liquid chromatography-tandem mass spectrometry. Prostaglandins Other Lipid Mediat. 2005 Dec;78(1-4):291-9. doi: 10.1016/j.prostaglandins.2005.10.001. Epub 2005 Nov 2. PMID 16303623
- [Background] Hardy G, Vergnaud S, Lunardi J, Peoc'h M, Bessard G, Stanke-Labesque F. 5-lipoxygenase expression and activity in aorta from streptozotocin-induced diabetic rats. Prostaglandins Other Lipid Mediat. 2005 Jan;75(1-4):91-103. doi: 10.1016/j.prostaglandins.2004.10.002. PMID 15789618
- [Background] Cipollone F, Mezzetti A, Fazia ML, Cuccurullo C, Iezzi A, Ucchino S, Spigonardo F, Bucci M, Cuccurullo F, Prescott SM, Stafforini DM. Association between 5-lipoxygenase expression and plaque instability in humans. Arterioscler Thromb Vasc Biol. 2005 Aug;25(8):1665-70. doi: 10.1161/01.ATV.0000172632.96987.2d. Epub 2005 Jun 2. PMID 15933245
- [Background] Dwyer JH, Allayee H, Dwyer KM, Fan J, Wu H, Mar R, Lusis AJ, Mehrabian M. Arachidonate 5-lipoxygenase promoter genotype, dietary arachidonic acid, and atherosclerosis. N Engl J Med. 2004 Jan 1;350(1):29-37. doi: 10.1056/NEJMoa025079. PMID 14702425
- [Background] Helgadottir A, Manolescu A, Thorleifsson G, Gretarsdottir S, Jonsdottir H, Thorsteinsdottir U, Samani NJ, Gudmundsson G, Grant SF, Thorgeirsson G, Sveinbjornsdottir S, Valdimarsson EM, Matthiasson SE, Johannsson H, Gudmundsdottir O, Gurney ME, Sainz J, Thorhallsdottir M, Andresdottir M, Frigge ML, Topol EJ, Kong A, Gudnason V, Hakonarson H, Gulcher JR, Stefansson K. The gene encoding 5-lipoxygenase activating protein confers risk of myocardial infarction and stroke. Nat Genet. 2004 Mar;36(3):233-9. doi: 10.1038/ng1311. Epub 2004 Feb 8. PMID 14770184
- [Derived] Boizel R, Bruttmann G, Benhamou PY, Halimi S, Stanke-Labesque F. Regulation of oxidative stress and inflammation by glycaemic control: evidence for reversible activation of the 5-lipoxygenase pathway in type 1, but not in type 2 diabetes. Diabetologia. 2010 Sep;53(9):2068-70. doi: 10.1007/s00125-010-1822-9. Epub 2010 Jun 10. No abstract available. PMID 20535444